CLINICAL TRIAL: NCT04503915
Title: A Multicenter Randomized Controlled Trial Comparing a Step-wise Increase Versus a Constant Dose of Estrogen Supplementation in Frozen-thawed Embryo Transfer Cycles Using Hormone Replacement
Brief Title: Estrogen Supplementation Mode in HRT-FET Cycle: a RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Haiyan Lin, Attending physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRT-E2
Record Dates: First submitted 2020-07-27; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Hormone Replacement Therapy; Estrogen; Live Birth Rate
Keywords: estrogen supplementation; HRT; Live birth rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constant group (Experimental): Women will receive oral estradiol valerate (Progynova®; Bayer Schering Pharma AG, Berlin, Germany) 3 mg bid for 14 days for endometrial priming from the second or third day of the menstrual cycle.
  Interventions: Procedure: different estrogen supplementation modes
- Step -up group (Active Comparator): Women will receive estradiol valerate 2mg once daily for 4 days from the second to fifth day,followed by 2mg bid for 4 days from the sixth to ninth day and then 3mg bid for 6 days from tenth to fifteenth day of menstrual cycle.
  Interventions: Procedure: different estrogen supplementation modes

INTERVENTIONS:
Procedure: different estrogen supplementation modes — The different estrogen supplementation modes are randomized into two groups.

SUMMARY:
A systematic review and meta-analysis concluded that there is insufficient evidence to recommend one particular protocol for HRT with regard to pregnancy rates after frozen embryo transfer, and no comparison of estrogen dose or route of administration was included in the review[7]. It is worth highlighting that the authors did not find any literature discussing the effect of estrogen dose and route of administration for HRT on reproductive outcomes. In 2016, a retrospective cohort study concluded that there is no difference in live birth rates between a constant dose versus an increasing dose of estrogen in oocyte donation cycles with oral or transdermal supplementation[6]. In order to provide good evidence about pattern of estrogen supplementation in HRT-FET, a randomized controlled study is urgently needed.

The present randomized controlled study aims to compare between a constant estrogen dose protocol and a step-wise increasing estrogen dose protocol on the live birth rate of HRT-FET cycles.

DETAILED DESCRIPTION:
The objective is to compare between a constant estrogen dose protocol and a step-wise increasing estrogen dose protocol on live birth rate of HRT-FET cycles.

This is a multicenter randomized controlled trial. Women undergoing HRT-FET will be recruited and randomized to use a constant estrogen dose protocol and a step-wise increasing estrogen dose protocol.

Participation in the study is totally voluntary. The subjects can withdraw from the study at any time and they will still receive standard medical care.

Women being scheduled for HRT-FET will be assessed for eligibility. Eligible women will be recruited in the study and each woman will only be included in the study once.

Informed written consent will be obtained prior to recruitment. The baseline characteristics will be collected. Transvaginal ultrasound will be done to measure the endometrial thickness on the day of progesterone supplementation. Embryo transfer will be performed 3 days or 5 days after progesterone use, depending on replacement of cleaving stage embryos or blastocysts respectively.

ELIGIBILITY:
Inclusion Criteria:

* Women aged <42 years at the time of HRT-FET
* Replacing 1-2 early cleavage embryos or blastocysts after thawing.

Exclusion Criteria:

* Preimplantation genetic testing(PGT)
* Use of donor oocytes
* Hydrosalpinx shown on pelvic scanning and not surgically treated such as tubal ligation or resection
* Severe uterine adhesion
* The endometrial thickness cannot reach 8mm in previous fresh cycles or HRT -FET cycles

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 784 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
live-birth rate per ET | Up to 12 months
  Live birth was defined as the delivery of at least one live born baby beyond 28 weeks of gestation.

SECONDARY OUTCOMES:
clinical pregnancy rate | Up to 6 months
  - clinical pregnancy: presence of intrauterine gestational sac on pelvic ultrasound at 6 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No
Until the completion of the study.